CLINICAL TRIAL: NCT04240197
Title: Reliability of Pressure Waveform Analysis to Determine Correct Epidural Catheter Placement; a Comparison Between Pressure Transducer and the CompuFlo® CathCheck™ System
Brief Title: Epidural Waveforms: Pressure Transducer vs CompuFlo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EESOA5
Record Dates: First submitted 2020-01-18; First posted 2020-01-27 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Pressure Transducer (Sham Comparator): Epidural pressure waveforms will be measured by using a standard invasive monitor pressure transducer
  Interventions: Device: CompuFlo
- CompuFlo (Active Comparator): Epidural pressure waveforms will be measured by using the CompuFlo Instrument
  Interventions: Device: CompuFlo

INTERVENTIONS:
Device: CompuFlo — The occurrence of epidural pulse waves with CompuFlo and with standard pressure trnsducer
  Other Names: Standard Pressure Transducer

SUMMARY:
The purpose of this single arm, open label study will be to compare and evaluate the sensitivity and specificity of CompuFlo to detect epidural pulse waveforms (EPW) to assess the correct placement of the catheter in the epidural space when compared to the standard pressure transducer.

DETAILED DESCRIPTION:
40 patients who had an epidural functioning catheter previously positioned for anesthesia or analgesia will be enrolled. After removing the epidural filter and after having zeroed the instrument, the investigator will connect in a random fashion sequence, a standard pressure transducer attached to a standard invasive blood pressure monitor or to the CompuFlo CathCheck instrument to observe and record the occurrence of epidural pulsatile waveform.

The investigator will also note and evaluate:

The volume of saline priming necessary to obtain the waveform The effects of patient's position on the occurrence and amplitude of epidural pulsatile waveform

ELIGIBILITY:
Inclusion Criteria:

* patients with an epidural lumbar catheter for anesthesia or analgesia

Exclusion Criteria:

* patients with malfunction or dislodgement of the epidural catheter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pulse Wave | up to 15 minutes
  Occurrence of epidural pulse wave

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Città di Roma Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hilber ND, Rijs K, Klimek M, Saenz G, Aloweidi A, Rossaint R, Heesen M. A systematic review of the diagnostic accuracy of epidural wave form analysis to identify the epidural space in surgical and labor patients. Minerva Anestesiol. 2019 Apr;85(4):393-400. doi: 10.23736/S0375-9393.18.13089-6. Epub 2018 Nov 22. PMID 30482001